CLINICAL TRIAL: NCT05424653
Title: To Evaluate Safety and Effectiveness of Transcatheter Aortic Valve System in Patients With Severe Symptomatic Aortic Insufficiency
Brief Title: To Evaluate Safety and Effectiveness of Transcatheter Aortic Valve System in Patients With Severe Aortic Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu Silara Meditech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Silara202101
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Aortic Insufficiency
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe Symptomatic Aortic Regurgitation (Experimental): Patients will be treated with transcatheter aortic valve system
  Interventions: Device: Transcatheter Aortic Valve System

INTERVENTIONS:
Device: Transcatheter Aortic Valve System — Procedure: Transcatheter Aortic Valve Replacement

SUMMARY:
To Evaluate the Safety and Effectiveness of Transcatheter Aortic Valve System ( Chengdu Silara Medtech Inc. ,Chengdu, China)in Patients with Severe Symptomatic Aortic Insufficiency

DETAILED DESCRIPTION:
Transcatheter Aortic Valve System (Chengdu Silara Medtech Inc. ,Chengdu, China) will be used for this study. To evaluate the feasibility , safety and effectiveness of Transcatheter aortic valve system.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years old;
2. Subjects with symptomatic severe aortic valve regurgitation.
3. NYHA Functional Class ≥II.
4. Life expectancy after aortic valve implantation thought to be >1 year，
5. Native valvular or peripheral vascular anatomy is appropriate for TAVR.
6. Patient is assessed by at least two cardiothoracic surgeons and recorded as not suitable for surgery (defined as a risk of operative mortality after 30 days>50%，or severe irreversible comorbidities or other factors affecting surgery (e.g., porcelain aorta, frailty, chest malformation, severe liver disease, severe lung disease, etc.)), or patients at high risk of surgery（Euroscore≥20%, or STS≥8）,or patient not agree open surgery.
7. Patient can understand the purpose of the study, voluntarily participates and signs the informed consent form and is willing to accept the relevant examination and clinical follow-up visits.

Exclusion Criteria:

1. Anatomy is not appropriate for percutaneous valve implantation. Native valve annulus diameter is not in the scope of application(native TAV diameter ≤20mm,or ≥28mm
2. Evidence of an acute myocardial infarction within 30 days prior to the study procedure, defined as: Q-wave myocardial infarction, or non-Q-wave myocardial infarction, with CK-MB≥ 2x normal and/or elevated Tn (WHO definition).
3. Any treatment for traumatic cardiac surgery within 30 day prior to the study procedure(except coronary revascularization).
4. Hematological abnormality, defined as: Leukopenia (WBC <3×109/L), acute anemia (Hb <90g/L), or thrombocytopenia (platelet count<50×109/L), history of bleeding diathesis or coagulopathy.
5. Severe ventricular insufficiency. Left ventricular ejection fraction (LVEF) <20%.
6. Echocardiographic evidence of intra-cardiac thrombus or vegetation etc.
7. Active pepticulcer or upper GI bleeding within 3 months prior to the study procedure.
8. Cerebral Vascular Accident (CVA) within 3 months prior to the study procedure,including TIA.
9. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine , clopidogrel and high polymer material, or sensitivity to contrast media, which cannot be adequately pre-medicated.
10. Patients with infective endocarditis or other active stage of infection. Currently participating in an investigational drug or another device trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Device success | Immediate post- procedure
  Device Success is defined as a composite of :
  Absence of procedural mortality AND Successful vascular access, delivery and deployment of the device, and successful retrieval of the delivery system AND Correct positioning of prosthetic heart valve into the proper anatomical location AND Intended performance of the prosthetic heart valve (mean aortic valve gradient<20 mmHg or peak velocity<3 m/s, and no moderate or more prosthetic valve regurgitation
Rate of Procedure success | Immediate post procedure
  Procedure Success is defined as no death, stroke, myocardial infarction and renal failure occurred within 72 hours after the operation on the basis of the final device success.
Rate of none or trace AR | 30 days
Rate of All cause mortality,including Cardiac death, non-cardiac death and unexplained death | 30 days
  Percentage of subjects who died from all causes in this population
Incidence of MACCE | 30 days
  MACCE includs death, stroke, MI, re-procedure, conduction disturbances and cardiac arrhythmias

SECONDARY OUTCOMES:
Delivery system performance | Immediate post-procedure
  Delivery System Performance wil be evaluated subjectively by the researchers participating in the operation, which is generally classified as excellent, good ,average and poor.
Retrieval system performance (if need) | Immediate post-procedure
  Retrieval System Performance wil be evaluated subjectively by the researchers participating in the operation, which is generally classified as excellent, good ,average and poor.
Exchange system evaluation | Immediate post-procedure
  Exchange Systerm Evaluation wil be evaluated subjectively by the researchers participating in the operation, which is generally classified as excellent, good ,average and poor.
Valvular function evaluation, including valve stenosis, AR, valve function(e.g. EOA, gradient) and PVL | Immediate post-procedure, 7 days or discharge, 30 days, 6 months and 12months
  The evaluation criteria refer to the 2012 edition of the Association for Valvular Academic Research (VARC-2) consensus document
Quality of Life Assessment | 30 days, 6 months,and 12 months
  SF-12
NYHA function | 7 days or discharge, 30 days, 6 months ,12 months
All-cause Mortality | Immediate post- procedure ,7 days /discharge, 6 months and 12 months
Rate of moderate to severe AR | immediate post- procedure ,7 days /discharge, 6 months and 12 months
Incidence of Myocardial Infarction | immediate post- procedure, 7 days /discharge, 30 days, 6 months and 12months
Incidence of MACCE | Immediate post- procedure, 7 days /discharge, 6 months and 12months.
  including death, stroke, MI, re-procedure, Conduction disturbances and cardiac arrhythmias
Incidence of Bleeding(life-threatening or disabling and major) | Immediate post- procedure, 7 days /discharge, 30 days, 6 months and 12 months
Incidence of stroke | 7 days /discharge, 30 days, 6 months and 12 months
Incidence of AKI | 7 days /discharge, 30 days, 6 months and 12 months
  including AKIN stage 2 and 3,or renal replacement therapy (RRT:Hemodialysis, abdomen Cavity dialysis, hemofiltration)
Incidence of Permanent Pacemaker Implantation | 7 days /discharge, 30 days, 6 months and 12 months
Incidence of major vascular complications | Immediate post- procedure, 7 days /discharge, 30 days, 6 months, 12 months
Incidence of Conduction disturbances and cardiac arrhythmias | Immediate post- procedure, 7 days /discharge, 30 days, 6 months, 12 months
Incidence of other TAVI-related complications | at immediate post- procedure, 7 days /discharge, 30 days, 6 months, 12 month
  including transfer to surgery , accidental heart-lung machine, coronary obstruction, ventricular septal rupture, mitral valve damage or dysfunction，cardiac tamponade，endocarditis ，valvular thrombus，valve migration(shifting, detachment, embolism, error deployment）,valve in valve

CONTACTS AND LOCATIONS:
Overall Officials: Jincheng Liu, Principal Investigator — The First Affiliated Hospital,the Air Force Medical University